CLINICAL TRIAL: NCT05180409
Title: The Prognostic Value of Simultaneous Assessment of Microcirculation Alteration With Sublingual Microcirculation and Near-infrared Spectroscopy on the Acute Respiratory Distress Syndrome of Various Phenotypes
Brief Title: Assessment of Microcirculation Alteration With Both Sublingual Microcirculation and Near-infrared Spectroscopy on ARDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMRPG3K2131
Record Dates: First submitted 2021-11-29; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-07

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Microcirculation; Near-infrared spectroscopy; Sublingual microcirculation; ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Microcirculatory alterations are frequently observed in critically ill and severe sepsis patients characterized by a decrease in capillary density and an increase in heterogeneity of perfusion. This derangements result in microcirculatory shunting and oxygen extraction deficit, and plays a major role in the pathophysiology of sepsis and multi-organ failure. Loss of hemodynamic coherence between the macro- and microcirculation results in persistent and incomplete reversal of microcirculatory and regional hypoxia that is the major factor contributing to the development of organ failure.

Current techniques permitting monitoring the microcirculation can be classified in two main groups: (1) Methods for evaluation of local tissue oxygenation as a surrogate of microcirculatory blood flow. (2)Methods allowing direct visualization of the microvascular network and microcirculatory blood flow.

Near-infrared spectroscopy (NIRS) is a non-invasive technique for evaluating tissue oxygenation in vessels with a diameter < 1 mm (arterioles, capillaries, and venules). Recent systemic review studies have showed that patients with severe sepsis or septic shock have lower levels of StO2, moreover, survivors present higher levels of StO2 compared with non-survivors. Reactive hyperemia during vascular occlusion test (VOT) can be considered an integral test of microcirculatory reactivity, evaluating the tissue's ability to adjust oxygen extraction capabilities to oxygen delivery after a hypoxic stimulus induced by a transient interruption in blood flow. Continuous StO2 measurement and VOT derived StO2 deoxygenation slope and StO2 recovery slope have been found to be predictors of mortality and organ dysfunction.

Sublingual microcirculation allows direct visualization of the sublingual microcirculation and for quantitative determination of variables of flow, capillary density, and flow distribution. Microvascular alterations including decreased functional capillary density, increased perfusion heterogeneity, and increased proportion of stopped and intermittently perfused capillaries, are more severe in non-survivors than in survivors. In addition, persistence of these alterations was strongly and independently correlated with multi-organ failure and mortality.

ARDS is the most severe form of acute lung injury in ICU with mortality about 45% without achievement in ten years. However, only few studies were focused on the microcirculatory alterations in ARDS patients.

DETAILED DESCRIPTION:
Microcirculation consists of a branching network of small blood vessels (<100 μm diameter) that includes the arterioles, capillaries, and venules, and plays a pivotal role in the delivery of oxygen to tissue cells. Microcirculatory alterations are frequently observed in critically ill patients, and especially in patients with severe sepsis. These alterations are characterized by a decrease in capillary density that determines an increase in the diffusion distance of oxygen to tissues and an increase in heterogeneity of perfusion. This microcirculatory derangements involve the consequent presence of under or not perfused capillaries in close proximity to well perfused capillaries. Therefore, these functionally vulnerable microcirculatory areas may become hypoxic, resulting in an oxygen extraction deficit. This phenomenon has been termed "microcirculatory shunting" and plays a major role in the pathophysiology of sepsis and multi-organ failure.

Persistent and incomplete reversal of microcirculatory and regional hypoxia is considered to be a major factor contributing to the development and maintenance of multiple organ failure. Unfortunately, alterations in microvascular perfusion often persist after the correction of systemic hemodynamic abnormalities, and their severity is associated with a poor outcome. Such a loss of hemodynamic coherence between the macro- and microcirculation has been described in several clinical and experimental studies and has been found to be an independent predictor of adverse outcome and organ dysfunction. The microcirculation has been suggested to be the motor of sepsis.

Conceptually, current techniques that permit monitoring the microcirculation can be classified in two main groups: (1) Methods that allow evaluation of local tissue oxygenation as a surrogate of microcirculatory blood flow. (2) Methods that allow direct visualization of the microvascular network and microcirculatory blood flow.

Near-infrared spectroscopy (NIRS) has been used as a tool to monitor tissue oxygen saturation (StO2) in acutely ill patients and has been proposed as a tool to quantify microvascular dysfunction in patients with sepsis. According to Beer's law, the NIRS signal is limited to vessels that have a diameter less than 1 mm (arterioles, capillaries, and venules), but, as 75% of the blood in a skeletal muscle is venous, NIRS StO2 measurements mostly represent local venous hemoglobin O2 saturation. NIRS has been used in different clinical conditions such as severe trauma, hemorrhagic shock, septic shock, and cardiogenic shock or severe cardiac failure. The utility of and application of NIRS in intensive care mainly involved three main NIRS measurements: (1) continuous tissue oxygen saturation (StO2) measurement; 2) StO2 deoxygenation slope (DecStO2 slope) in response to vascular occlusion test (VOT test); and 3) StO2 recovery slope (RincStO2 slope) in response to VOT.

Tissue oxygen saturation (StO2) has been proposed as a marker of tissue perfusion depending on the device used and the location of the measurement. A systemic review and mea-analysis had showed that patients with severe sepsis or septic shock have lower levels of StO2, and RincStO2 slope. Moreover, survivors from severe sepsis or septic shock present higher levels of StO2 and RincStO2 compared with non-survivors. The VOT is a provocative test in which StO2 is measured on a distal site (such as the thenar eminence or forearm) whilst a transient rapid vascular occlusion is performed, using a sphygmomanometer, for either a defined time interval (for example, 3 minutes) or until the StO2 decreases to a defined minimal threshold. The ischemic tissue then induces vasodilation of surrounding arterioles, metarterioles and pre-capillary sphincters to decrease local vascular resistance and regain blood flow. Once this threshold is reached, the tourniquet is released and blood flow is restored. There is a reactive hyperemic response which represents the tissue's ability to auto-regulate blood flow and oxygenation. Several parameters arise from this technique, including: 1. the rate of deoxygenation (RdecStO2), thought to reflect the local metabolic rate, 2. the rate of reoxygenation (RincStO2), thought to reflects the time required to wash out stagnant blood and is thought to be determined by local cardiovascular reserve and microcirculatory flow, and the post-obstructive hyperemic response.

For the rate of StO2 increase (RincStO2), or termed StO2 recovery slope, it is assumed that when the StO2 recovery slope is reduced, the capacities of recruiting microvessels in response to a hypoxic stimulus are lower. Many papers have demonstrated that the RincStO2 is decreased in septic patients. The StO2 recovery slope had been shown to be lower in septic patients and that the presence of this alteration in the first 24 h of sepsis and its persistence were associated with a worse outcome. Among the septic patients, the RincStO2 was higher in survivors than in non-survivors and was most strongly associated with organ dysfunction and mortality.

However, StO2 is not a direct measurement of microvascular blood flow, but an index of tissue oxygenation which is dependent on the balance between O2 delivery (DO2) and oxygen consumption (VO2). Any change in StO2 can reflect a change in flow in the same direction and/or a change in metabolism in the opposite direction. More importantly, proportional changes in flow and metabolism may be associated with unchanged StO2. The vasoreactivity test evaluates microvascular reserve more than actual microvascular perfusion. Indeed, even though StO2 is slightly lower in septic patients compared to healthy volunteers, there is a huge overlap between the groups. No significant difference in StO2 between injured patients and healthy volunteers has been found among septic shock, post-surgery, and healthy subjects; between septic shock and normal volunteers; and between trauma patients and healthy subjects, or even higher tissue oxygen tension in patients with sepsis has been reported.

As a consequence, a vascular occlusion test (VOT) combined with StO2 measurement has been proposed to enhance the discriminatory power and to better evaluate the tissue micro-oxygenation in septic shock. The use of VOT has been shown to improve and expand the predictive ability of StO2 to scenarios such as trauma, severe sepsis and septic shock.

Micro-videoscopic techniques are assumed to be the gold standard for the study of the microcirculation as these allow the direct visualization of microvascular perfusion and characterization of its alterations. Recently, a third-generation lightweight handheld vital microscopes (CytoCam) was developed based on incident dark field imaging. Direct visualization of the sublingual microcirculation allows quantitative determination of capillary density, microvessel morphology, and dynamics of microcirculatory blood flow.

Variables of flow including Microvascular Flow Index (MFI) and proportion of perfused vessels (PPV), as well as capillary density including total vessel density (TVD) and perfused vessel density (PVD), and flow distribution Heterogeneity Index (HI) were calculated according to international criteria. The alterations seen in sepsis are often characterized by a highly heterogeneous perfusion, with stopped flow capillaries next to vessels with flowing cells.

Microvascular alterations, which are characterized by decreased functional capillary density, increased perfusion heterogeneity, and increased proportion of stopped and intermittently perfused capillaries, contribute to the defect in oxygen extraction observed in sepsis, and may be involved in the development of organ failure. Microcirculatory alterations are more severe in non-survivors than in survivors. The survival rate progressively decreased with quartiles of severity in alteration of the microcirculation. In addition, alterations in microvascular perfusion were one of the strongest predictors of outcome and remained independently associated with outcome in multivariate analysis. The time course of microvascular alterations also differs between survivors and non-survivors. Microvascular alterations improved over time in response to therapy in survivors but not in non-survivors. Conversely, the persistence of these microcirculatory alterations after the first 24 h was strongly and independently correlated with mortality secondary to circulatory failure in the early phase and to multi-organ failure in the late phase. For the flow parameter, in 2009, an international multicenter observational prevalence study in ICU patients involving 36 ICUs worldwide enrolling 501 patients identified microcirculatory alterations MFI < 2.6 in combination with tachycardia (heart rate > 90) as an independent risk factor for increased hospital mortality.

Among microcirculatory variables, there is no clear consensus on which microcirculatory perfusion parameter is most important. The decreased microcirculatory perfusion as measured by PPV, PVD, and MFI was associated with mortality. They reported that the PPV parameter was the strongest predictor of mortality and that this association was maintained in multiple logistic regression models for both early (< 24 h) and late (≥ 24 h) time points. In a similar study, impaired flow and increased heterogeneity of flow were significantly disturbed features of the microcirculation in non-survivors compared with survivors. Furthermore, in a study of 49 ICU patients in septic shock, there was no difference in microcirculatory perfusion parameters at the onset of shock, but survivors were able to restore their microcirculatory perfusion as indicated by significant differences in PPV. However, in the ProCESS trial, the measures of density, namely TVD, PVD, and De Backer score (an estimate of total density), to be associated with mortality at all time-points in a single model and at the 72-h time period. Therefore, which microcirculatory parameters having the most significant pathophysiologic impact still await for further studies to delineate.

Acute respiratory distress syndrome (ARDS) is the most severe form of acute lung injury in ICU. The hallmark of ARDS pathogenesis is marked increased permeability from endothelial and epithelial injury [58]. Persistent and marked tissue hypoxia and multiple organ failure are the main cause of death. The attributable mortality of ARDS remains high without achievement within the recent ten years. Recently, The Large Observational Study to Understand the Global Impact of Severe Acute Respiratory Failure (LUNG SAFE) study revealed that in the 29 144 patients admitted to participating ICUs, the hospital mortality was 34.9% for those with mild, 40.3% for moderate, and 46.1% for severe ARDS.

Therefore, from the aforementioned discussion for the two major assessment NIRS and sublingual microcirculation, the aims of our study are the followings:

1. To compare the predictive power of the NIRS and sublingual microcirculation for the prognosis of ARDS. Furthermore, whether the prognosis of ARDS can be predicted more precisely if investigators simultaneously assessing microcirculatory alteration with NIRS and sublingual microcirculation?
2. To delineate which parameters of microcirculatory alteration, variables of flow or density have the most significant pathophysiologic impact for the prognosis of ARDS?

ELIGIBILITY:
Inclusion Criteria:

* ARDS patients conforming to the Berlin Definition of Acute Respiratory Distress Syndrome
* ventilatory support with mechanical ventilation

Exclusion Criteria:

* age < 18 years
* pregnancy
* established "Do Not Resuscitate" orders prior to enrollment
* acute cerebrovascular event (primary diagnosis)
* combined with acute coronary syndrome with myocardial infarction (primary diagnosis)
* acute and active gastrointestinal bleeding (primary diagnosis)
* requirement for immediate surgery
* inability to obtain written informed consent

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: admitted to medical ICU and the hemodynamics is stable (mean arterial pressure MAP > 60 mmHg with no change in vasopressor infusion rate for 2 hours) will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Predictive power of the near-infrared spectroscopy and sublingual microcirculation for the prognosis of ARDS | 28 days mortality after admission into ICU
  The outcomes variables planned to be recorded are area under the receiver operating characteristic (ROC) curve for the sublingual microcirculation and near-infrared spectroscopy to predict mortality of ARDS

CONTACTS AND LOCATIONS:
Overall Officials: Chung Chi Huang, MD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ince C. The rationale for microcirculatory guided fluid therapy. Curr Opin Crit Care. 2014 Jun;20(3):301-8. doi: 10.1097/MCC.0000000000000091. PMID 24758985
- [Result] De Backer D, Ospina-Tascon G, Salgado D, Favory R, Creteur J, Vincent JL. Monitoring the microcirculation in the critically ill patient: current methods and future approaches. Intensive Care Med. 2010 Nov;36(11):1813-25. doi: 10.1007/s00134-010-2005-3. Epub 2010 Aug 6. PMID 20689916
- [Result] Goldman D, Bateman RM, Ellis CG. Effect of decreased O2 supply on skeletal muscle oxygenation and O2 consumption during sepsis: role of heterogeneous capillary spacing and blood flow. Am J Physiol Heart Circ Physiol. 2006 Jun;290(6):H2277-85. doi: 10.1152/ajpheart.00547.2005. Epub 2006 Jan 6. PMID 16399873
- [Result] Ince C. The microcirculation is the motor of sepsis. Crit Care. 2005;9 Suppl 4(Suppl 4):S13-9. doi: 10.1186/cc3753. Epub 2005 Aug 25. PMID 16168069
- [Result] Gruartmoner G, Mesquida J, Ince C. Microcirculatory monitoring in septic patients: Where do we stand? Med Intensiva. 2017 Jan-Feb;41(1):44-52. doi: 10.1016/j.medin.2016.11.011. Epub 2017 Jan 17. English, Spanish. PMID 28104277
- [Result] Vincent JL, De Backer D. Microvascular dysfunction as a cause of organ dysfunction in severe sepsis. Crit Care. 2005;9 Suppl 4(Suppl 4):S9-12. doi: 10.1186/cc3748. Epub 2005 Aug 25. PMID 16168075
- [Result] De Backer D, Creteur J, Preiser JC, Dubois MJ, Vincent JL. Microvascular blood flow is altered in patients with sepsis. Am J Respir Crit Care Med. 2002 Jul 1;166(1):98-104. doi: 10.1164/rccm.200109-016oc. PMID 12091178
- [Result] De Backer D, Donadello K, Sakr Y, Ospina-Tascon G, Salgado D, Scolletta S, Vincent JL. Microcirculatory alterations in patients with severe sepsis: impact of time of assessment and relationship with outcome. Crit Care Med. 2013 Mar;41(3):791-9. doi: 10.1097/CCM.0b013e3182742e8b. PMID 23318492
- [Result] Sakr Y, Dubois MJ, De Backer D, Creteur J, Vincent JL. Persistent microcirculatory alterations are associated with organ failure and death in patients with septic shock. Crit Care Med. 2004 Sep;32(9):1825-31. doi: 10.1097/01.ccm.0000138558.16257.3f. PMID 15343008
- [Result] Shapiro NI, Arnold R, Sherwin R, O'Connor J, Najarro G, Singh S, Lundy D, Nelson T, Trzeciak SW, Jones AE; Emergency Medicine Shock Research Network (EMShockNet). The association of near-infrared spectroscopy-derived tissue oxygenation measurements with sepsis syndromes, organ dysfunction and mortality in emergency department patients with sepsis. Crit Care. 2011;15(5):R223. doi: 10.1186/cc10463. Epub 2011 Sep 22. PMID 21939529
- [Result] Hernandez G, Boerma EC, Dubin A, Bruhn A, Koopmans M, Edul VK, Ruiz C, Castro R, Pozo MO, Pedreros C, Veas E, Fuentealba A, Kattan E, Rovegno M, Ince C. Severe abnormalities in microvascular perfused vessel density are associated to organ dysfunctions and mortality and can be predicted by hyperlactatemia and norepinephrine requirements in septic shock patients. J Crit Care. 2013 Aug;28(4):538.e9-14. doi: 10.1016/j.jcrc.2012.11.022. Epub 2013 Apr 6. PMID 23566729
- [Result] Meinders AJ, Nieuwenhuis L, Ince C, Bos WJ, Elbers PW. Haemodialysis Impairs the Human Microcirculation Independent from Macrohemodynamic Parameters. Blood Purif. 2015;40(1):38-44. doi: 10.1159/000380902. Epub 2015 Jun 11. PMID 26068109
- [Result] Ince C. Hemodynamic coherence and the rationale for monitoring the microcirculation. Crit Care. 2015;19 Suppl 3(Suppl 3):S8. doi: 10.1186/cc14726. Epub 2015 Dec 18. PMID 26729241
- [Result] Pranskunas A, Koopmans M, Koetsier PM, Pilvinis V, Boerma EC. Microcirculatory blood flow as a tool to select ICU patients eligible for fluid therapy. Intensive Care Med. 2013 Apr;39(4):612-9. doi: 10.1007/s00134-012-2793-8. Epub 2012 Dec 20. PMID 23263029
- [Result] Hanson JP, Lam SW, Mohanty S, Alam S, Pattnaik R, Mahanta KC, Hasan MU, Charunwatthana P, Mishra SK, Day NP, White NJ, Dondorp AM. Fluid resuscitation of adults with severe falciparum malaria: effects on Acid-base status, renal function, and extravascular lung water. Crit Care Med. 2013 Apr;41(4):972-81. doi: 10.1097/CCM.0b013e31827466d2. PMID 23324951
- [Result] Jhanji S, Stirling S, Patel N, Hinds CJ, Pearse RM. The effect of increasing doses of norepinephrine on tissue oxygenation and microvascular flow in patients with septic shock. Crit Care Med. 2009 Jun;37(6):1961-6. doi: 10.1097/CCM.0b013e3181a00a1c. PMID 19384212
- [Result] Dubin A, Pozo MO, Casabella CA, Palizas F Jr, Murias G, Moseinco MC, Kanoore Edul VS, Palizas F, Estenssoro E, Ince C. Increasing arterial blood pressure with norepinephrine does not improve microcirculatory blood flow: a prospective study. Crit Care. 2009;13(3):R92. doi: 10.1186/cc7922. Epub 2009 Jun 17. PMID 19534818
- [Result] Buijs EA, Reiss IK, Kraemer U, Andrinopoulou ER, Zwiers AJ, Ince C, Tibboel D. Increasing mean arterial blood pressure and heart rate with catecholaminergic drugs does not improve the microcirculation in children with congenital diaphragmatic hernia: a prospective cohort study. Pediatr Crit Care Med. 2014 May;15(4):343-54. doi: 10.1097/PCC.0000000000000105. PMID 24622167
- [Result] Vincent JL, Taccone FS. Microvascular monitoring - Do 'global' markers help? Best Pract Res Clin Anaesthesiol. 2016 Dec;30(4):399-405. doi: 10.1016/j.bpa.2016.10.006. Epub 2016 Nov 3. PMID 27931643
- [Result] Arnold RC, Dellinger RP, Parrillo JE, Chansky ME, Lotano VE, McCoy JV, Jones AE, Shapiro NI, Hollenberg SM, Trzeciak S. Discordance between microcirculatory alterations and arterial pressure in patients with hemodynamic instability. J Crit Care. 2012 Oct;27(5):531.e1-7. doi: 10.1016/j.jcrc.2012.02.007. Epub 2012 May 15. PMID 22591569
- [Result] Ince C, Sinaasappel M. Microcirculatory oxygenation and shunting in sepsis and shock. Crit Care Med. 1999 Jul;27(7):1369-77. doi: 10.1097/00003246-199907000-00031. PMID 10446833
- [Result] Top AP, Ince C, de Meij N, van Dijk M, Tibboel D. Persistent low microcirculatory vessel density in nonsurvivors of sepsis in pediatric intensive care. Crit Care Med. 2011 Jan;39(1):8-13. doi: 10.1097/CCM.0b013e3181fb7994. PMID 21076287
- [Result] Edul VS, Enrico C, Laviolle B, Vazquez AR, Ince C, Dubin A. Quantitative assessment of the microcirculation in healthy volunteers and in patients with septic shock. Crit Care Med. 2012 May;40(5):1443-8. doi: 10.1097/CCM.0b013e31823dae59. PMID 22430243
- [Result] Trzeciak S, McCoy JV, Phillip Dellinger R, Arnold RC, Rizzuto M, Abate NL, Shapiro NI, Parrillo JE, Hollenberg SM; Microcirculatory Alterations in Resuscitation and Shock (MARS) investigators. Early increases in microcirculatory perfusion during protocol-directed resuscitation are associated with reduced multi-organ failure at 24 h in patients with sepsis. Intensive Care Med. 2008 Dec;34(12):2210-7. doi: 10.1007/s00134-008-1193-6. Epub 2008 Jul 2. PMID 18594793
- [Result] Creteur J. Muscle StO2 in critically ill patients. Curr Opin Crit Care. 2008 Jun;14(3):361-6. doi: 10.1097/MCC.0b013e3282fad4e1. PMID 18467900
- [Result] De Blasi RA, Palmisani S, Alampi D, Mercieri M, Romano R, Collini S, Pinto G. Microvascular dysfunction and skeletal muscle oxygenation assessed by phase-modulation near-infrared spectroscopy in patients with septic shock. Intensive Care Med. 2005 Dec;31(12):1661-8. doi: 10.1007/s00134-005-2822-y. Epub 2005 Oct 5. PMID 16205889
- [Result] Gomez H, Torres A, Polanco P, Kim HK, Zenker S, Puyana JC, Pinsky MR. Use of non-invasive NIRS during a vascular occlusion test to assess dynamic tissue O(2) saturation response. Intensive Care Med. 2008 Sep;34(9):1600-7. doi: 10.1007/s00134-008-1145-1. Epub 2008 Jun 4. PMID 18523754
- [Result] Beilman GJ, Groehler KE, Lazaron V, Ortner JP. Near-infrared spectroscopy measurement of regional tissue oxyhemoglobin saturation during hemorrhagic shock. Shock. 1999 Sep;12(3):196-200. doi: 10.1097/00024382-199909000-00005. PMID 10485597
- [Result] Taylor JH, Mulier KE, Myers DE, Beilman GJ. Use of near-infrared spectroscopy in early determination of irreversible hemorrhagic shock. J Trauma. 2005 Jun;58(6):1119-25. doi: 10.1097/01.ta.0000169951.20802.20. PMID 15995457
- [Result] Podbregar M, Mozina H. Skeletal muscle oxygen saturation does not estimate mixed venous oxygen saturation in patients with severe left heart failure and additional severe sepsis or septic shock. Crit Care. 2007;11(1):R6. doi: 10.1186/cc5153. PMID 17227587
- [Result] Pareznik R, Knezevic R, Voga G, Podbregar M. Changes in muscle tissue oxygenation during stagnant ischemia in septic patients. Intensive Care Med. 2006 Jan;32(1):87-92. doi: 10.1007/s00134-005-2841-8. Epub 2005 Nov 1. PMID 16261341
- [Result] Doerschug KC, Delsing AS, Schmidt GA, Haynes WG. Impairments in microvascular reactivity are related to organ failure in human sepsis. Am J Physiol Heart Circ Physiol. 2007 Aug;293(2):H1065-71. doi: 10.1152/ajpheart.01237.2006. Epub 2007 May 4. PMID 17483235
- [Result] Skarda DE, Mulier KE, Myers DE, Taylor JH, Beilman GJ. Dynamic near-infrared spectroscopy measurements in patients with severe sepsis. Shock. 2007 Apr;27(4):348-53. doi: 10.1097/01.shk.0000239779.25775.e4. PMID 17414414
- [Result] Creteur J, Carollo T, Soldati G, Buchele G, De Backer D, Vincent JL. The prognostic value of muscle StO2 in septic patients. Intensive Care Med. 2007 Sep;33(9):1549-56. doi: 10.1007/s00134-007-0739-3. Epub 2007 Jun 16. PMID 17572876
- [Result] 36. Matsushita K, Homma S, Okada E. Influence of adipose tissue on muscle oxygenation measurement with NIRS instrument. Proc SPIE. 1998; 2194:159 -165
- [Result] Bezemer R, Lima A, Myers D, Klijn E, Heger M, Goedhart PT, Bakker J, Ince C. Assessment of tissue oxygen saturation during a vascular occlusion test using near-infrared spectroscopy: the role of probe spacing and measurement site studied in healthy volunteers. Crit Care. 2009;13 Suppl 5(Suppl 5):S4. doi: 10.1186/cc8002. Epub 2009 Nov 30. PMID 19951388
- [Result] 38. Bhutta A, Fontenot E, Ford J, et al. The use of non-invasive cerebral oximeter as a surrogate for mixed venous saturations in children. Crit Care Med. 2004; 32:12-24
- [Result] Bhatia A, Gupta AK. Neuromonitoring in the intensive care unit. II. Cerebral oxygenation monitoring and microdialysis. Intensive Care Med. 2007 Aug;33(8):1322-8. doi: 10.1007/s00134-007-0660-9. Epub 2007 May 24. PMID 17522846
- [Result] Greisen G. Is near-infrared spectroscopy living up to its promises? Semin Fetal Neonatal Med. 2006 Dec;11(6):498-502. doi: 10.1016/j.siny.2006.07.010. Epub 2006 Sep 7. PMID 16959556
- [Result] Gagnon RE, Macnab AJ, Gagnon FA, Blackstock D, LeBlanc JG. Comparison of two spatially resolved NIRS oxygenation indices. J Clin Monit Comput. 2002 Dec;17(7-8):385-91. doi: 10.1023/a:1026274124837. PMID 14650633
- [Result] Yoshitani K, Kawaguchi M, Tatsumi K, Kitaguchi K, Furuya H. A comparison of the INVOS 4100 and the NIRO 300 near-infrared spectrophotometers. Anesth Analg. 2002 Mar;94(3):586-90; table of contents. doi: 10.1097/00000539-200203000-00020. PMID 11867380
- [Result] Owen-Reece H, Smith M, Elwell CE, Goldstone JC. Near infrared spectroscopy. Br J Anaesth. 1999 Mar;82(3):418-26. doi: 10.1093/bja/82.3.418. No abstract available. PMID 10434827
- [Result] Neto AS, Pereira VG, Manetta JA, Esposito DC, Schultz MJ. Association between static and dynamic thenar near-infrared spectroscopy and mortality in patients with sepsis: a systematic review and meta-analysis. J Trauma Acute Care Surg. 2014 Jan;76(1):226-33. doi: 10.1097/TA.0b013e3182a9221f. PMID 24368385
- [Result] Mulier KE, Skarda DE, Taylor JH, Myers DE, McGraw MK, Gallea BL, Beilman GJ. Near-infrared spectroscopy in patients with severe sepsis: correlation with invasive hemodynamic measurements. Surg Infect (Larchmt). 2008 Oct;9(5):515-9. doi: 10.1089/sur.2007.091. PMID 18687043
- [Result] Sair M, Etherington PJ, Peter Winlove C, Evans TW. Tissue oxygenation and perfusion in patients with systemic sepsis. Crit Care Med. 2001 Jul;29(7):1343-9. doi: 10.1097/00003246-200107000-00008. PMID 11445683
- [Result] Sherman H, Klausner S, Cook WA. Incident dark-field illumination: a new method for microcirculatory study. Angiology. 1971 May;22(5):295-303. doi: 10.1177/000331977102200507. No abstract available. PMID 5089888
- [Result] Aykut G, Veenstra G, Scorcella C, Ince C, Boerma C. Cytocam-IDF (incident dark field illumination) imaging for bedside monitoring of the microcirculation. Intensive Care Med Exp. 2015 Dec;3(1):40. doi: 10.1186/s40635-015-0040-7. Epub 2015 Jan 31. PMID 26215807
- [Result] Ince C, Boerma EC, Cecconi M, De Backer D, Shapiro NI, Duranteau J, Pinsky MR, Artigas A, Teboul JL, Reiss IKM, Aldecoa C, Hutchings SD, Donati A, Maggiorini M, Taccone FS, Hernandez G, Payen D, Tibboel D, Martin DS, Zarbock A, Monnet X, Dubin A, Bakker J, Vincent JL, Scheeren TWL; Cardiovascular Dynamics Section of the ESICM. Second consensus on the assessment of sublingual microcirculation in critically ill patients: results from a task force of the European Society of Intensive Care Medicine. Intensive Care Med. 2018 Mar;44(3):281-299. doi: 10.1007/s00134-018-5070-7. Epub 2018 Feb 6. PMID 29411044
- [Result] De Backer D, Hollenberg S, Boerma C, Goedhart P, Buchele G, Ospina-Tascon G, Dobbe I, Ince C. How to evaluate the microcirculation: report of a round table conference. Crit Care. 2007;11(5):R101. doi: 10.1186/cc6118. PMID 17845716
- [Result] Boerma EC, Mathura KR, van der Voort PH, Spronk PE, Ince C. Quantifying bedside-derived imaging of microcirculatory abnormalities in septic patients: a prospective validation study. Crit Care. 2005;9(6):R601-6. doi: 10.1186/cc3809. Epub 2005 Sep 22. PMID 16280059
- [Result] Spronk PE, Ince C, Gardien MJ, Mathura KR, Oudemans-van Straaten HM, Zandstra DF. Nitroglycerin in septic shock after intravascular volume resuscitation. Lancet. 2002 Nov 2;360(9343):1395-6. doi: 10.1016/s0140-6736(02)11393-6. PMID 12423989
- [Result] Vellinga NA, Boerma EC, Koopmans M, Donati A, Dubin A, Shapiro NI, Pearse RM, Machado FR, Fries M, Akarsu-Ayazoglu T, Pranskunas A, Hollenberg S, Balestra G, van Iterson M, van der Voort PH, Sadaka F, Minto G, Aypar U, Hurtado FJ, Martinelli G, Payen D, van Haren F, Holley A, Pattnaik R, Gomez H, Mehta RL, Rodriguez AH, Ruiz C, Canales HS, Duranteau J, Spronk PE, Jhanji S, Hubble S, Chierego M, Jung C, Martin D, Sorbara C, Tijssen JG, Bakker J, Ince C; microSOAP Study Group. International study on microcirculatory shock occurrence in acutely ill patients. Crit Care Med. 2015 Jan;43(1):48-56. doi: 10.1097/CCM.0000000000000553. PMID 25126880
- [Result] Farquhar I, Martin CM, Lam C, Potter R, Ellis CG, Sibbald WJ. Decreased capillary density in vivo in bowel mucosa of rats with normotensive sepsis. J Surg Res. 1996 Feb 15;61(1):190-6. doi: 10.1006/jsre.1996.0103. PMID 8769965
- [Result] Ellis CG, Bateman RM, Sharpe MD, Sibbald WJ, Gill R. Effect of a maldistribution of microvascular blood flow on capillary O(2) extraction in sepsis. Am J Physiol Heart Circ Physiol. 2002 Jan;282(1):H156-64. doi: 10.1152/ajpheart.2002.282.1.H156. PMID 11748059
- [Result] Massey MJ, Hou PC, Filbin M, Wang H, Ngo L, Huang DT, Aird WC, Novack V, Trzeciak S, Yealy DM, Kellum JA, Angus DC, Shapiro NI; ProCESS investigators. Microcirculatory perfusion disturbances in septic shock: results from the ProCESS trial. Crit Care. 2018 Nov 20;22(1):308. doi: 10.1186/s13054-018-2240-5. PMID 30458880
- [Result] Ware LB, Matthay MA. The acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1334-49. doi: 10.1056/NEJM200005043421806. No abstract available. PMID 10793167
- [Result] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337